CLINICAL TRIAL: NCT00271024
Title: Efficacy of Naltrexone in Women's Smoking Cessation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 13976A (R01 DA016834); R01DA016834 (NIH)
Record Dates: First submitted 2005-12-28; First posted 2005-12-29 (Estimated); Results first posted 2013-04-26 (Estimated); Last update posted 2023-03-23 (Actual); Status verified 2023-02

CONDITIONS: Smoking; Smoking Cessation
Keywords: Smoking; Smoking Cessation
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Naltrexone; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Male Naltrexone (Experimental): 50 mg Naltrexone tablet
  Interventions: Drug: Naltrexone (drug)
- Female Naltrexone (Experimental): Females receiving either naltrexone (50 mg)
  Interventions: Drug: Naltrexone (drug)
- Male Placebo (Placebo Comparator): Males receiving Placebo (sugar pill)
  Interventions: Drug: Placebo (for Naltrexone)
- Female Placebo (Placebo Comparator): Females receiving placebo (sugar pill)
  Interventions: Drug: Placebo (for Naltrexone)

INTERVENTIONS:
Drug: Naltrexone (drug) — 50 mg q.d. for 13 weeks
  Arms: Female Naltrexone; Male Naltrexone
Drug: Placebo (for Naltrexone) — Sugar pill manufactured to mimic Naltrexone tablet
  Arms: Female Placebo; Male Placebo

SUMMARY:
The purpose of the proposed study is to conduct a randomized, double-blind clinical trial to compare adjunct treatment with 50 mg oral naltrexone vs. placebo in conjunction with standard smoking cessation treatment with nicotine patch and counseling.

Hypotheses:

1. Naltrexone will improve smoking cessation quit rates, as measured at the end of active treatment (3 months) and during long term follow up (1 year).
2. Weight and smoking-related variables (i.e., less weight gain, as well as reduced craving and withdrawal) will be important factors by which naltrexone improves smoking cessation outcome.
3. These effects are predicted to be stronger in women compared to men.

DETAILED DESCRIPTION:
Although women may be particularly susceptible to the damaging effects of chronic cigarette smoking, evidence indicates that they may have more difficulty in maintaining smoking cessation than men. Given women's reduced response to nicotine replacement and other traditional treatments to habitual cigarette smoking, more targeted pharmacotherapy and intervention strategies may be necessary to improve their quit rates. Preliminary data by our group and others indicate that the opioid antagonist naltrexone may be an effective adjunctive pharmacotherapy approach for female smokers. The purpose of the proposed study is to conduct a randomized clinical trial to compare adjunct treatment with 50 mg oral naltrexone vs. placebo in conjunction with standard smoking cessation treatment with nicotine patch and counseling. Participants (N=324) will be randomized to receive either naltrexone or placebo starting one week prior to the quit date (25 mg for three days; 50 mg thereafter) and continue for 12 weeks after the quit date. The effects of naltrexone will be evaluated during the pre-quit date period, initial smoking cessation, relapse prevention, and at one year follow-up. It is hypothesized that sex will moderate the effects of naltrexone on outcome, with naltrexone improving prolonged abstinence quit rates in women but not in men. The secondary goal will be to elucidate the mechanism underlying women's treatment response to naltrexone. Weight (relative weight gain and weight concerns) and smoking-related variables (reduced cigarette pleasure, taste, craving and relief of negative withdrawal affect) may be important factors by which naltrexone improves quit rates in women. Medication compliance, psychosocial stress and levels of naltrexone's metabolite, 6-B-naltrexol, will also be examined. In sum, the proposed clinical trial will provide a comprehensive study of sex differences in response to adjunct treatment with naltrexone for smoking cessation. Given the public health concerns and significant health consequences of women's continued high rates of smoking, the proposed study may provide important information on a novel treatment strategy targeting the endogenous opioid system to selectively aid in women's smoking cessation.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65, male or female
2. Cigarette smoker of at least 15 but no more than 40 cigarettes daily for at least two years
3. Current diagnosis of DSM-IV Nicotine Dependence, based on SCID interview
4. Relatively healthy, with no medical or psychiatric conditions that would adversely interact with study parameters (see exclusion criteria for specific details)
5. Desire to quit smoking (self-report rating of interest in quitting at least a 7 on a 10-point scale)
6. Nicometer® cotinine level at baseline at least a 5 on a 6-point scale
7. Reports not quitting smoking in the past three months for more than one week duration
8. Agrees to attend behavioral counseling sessions and complete study measures
9. Has stable residence and telephone and can provide the name of an outside household collateral family member or close friend

Exclusion Criteria:

1. Substance Dependence in the last one year (other than DSM-IV Nicotine Dependence) or any history of Opioid Dependence (lifetime)
2. Major psychiatric disorder in the last one year, including Axis I disorders or any history of moderate/severe Axis II Disorder, Bipolar Disorder or Psychotic Disorder, based on SCID interview and standard cut-off thresholds on screening questionnaires
3. Past or current medical disorders (cardiovascular, hepatic, neurological, endocrine, etc.) which may adversely interact with study measures
4. Clinically significant lab test abnormalities, positive urine toxicology, or positive pregnancy test
5. Currently pregnant, plans to become pregnant, or lack of effective birth control over next three months, and/or currently lactating, or plans for breastfeeding over next three months
6. History of adverse reaction to opioid antagonist or nicotine replacement treatment
7. Use of any medication that may adversely interact with study measures (antidepressants, phenothiazines, benzodiazepines, etc.); recent or regular use of an opioid medication
8. Unwillingness to attend smoking cessation treatment sessions, take the nicotine patch, or be randomized into medication or placebo conditions, or be available for follow-up assessments
9. Unwillingness to agree to DNA analysis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 333 (Actual)
Dates: Start 2005-12; Primary Completion 2009-06 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C King, PhD, Principal Investigator — The University of Chicago, Department of Psychiatry
Locations (1):
- The University of Chicago, Department of Psychiatry, Chicago, Illinois, United States

REFERENCES:
- [Background] King AC, Meyer PJ. Naltrexone alteration of acute smoking response in nicotine-dependent subjects. Pharmacol Biochem Behav. 2000 Jul;66(3):563-72. doi: 10.1016/s0091-3057(00)00258-6. PMID 10899371
- [Background] King AC. Role of naltrexone in initial smoking cessation: preliminary findings. Alcohol Clin Exp Res. 2002 Dec;26(12):1942-4. doi: 10.1097/01.ALC.0000041003.44118.9B. No abstract available. PMID 12500129
- [Background] Epstein AM, King AC. Naltrexone attenuates acute cigarette smoking behavior. Pharmacol Biochem Behav. 2004 Jan;77(1):29-37. doi: 10.1016/j.pbb.2003.09.017. PMID 14724039
- [Background] King A, de Wit H, Riley RC, Cao D, Niaura R, Hatsukami D. Efficacy of naltrexone in smoking cessation: a preliminary study and an examination of sex differences. Nicotine Tob Res. 2006 Oct;8(5):671-82. doi: 10.1080/14622200600789767. PMID 17008194
- [Derived] King AC, Cao D, Zhang L, O'Malley SS. Naltrexone reduction of long-term smoking cessation weight gain in women but not men: a randomized controlled trial. Biol Psychiatry. 2013 May 1;73(9):924-30. doi: 10.1016/j.biopsych.2012.09.025. Epub 2012 Nov 22. PMID 23177384
- See also: Main Study Website — http://stopsmoking.uchicago.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment for this study lasted from August 2006-March 2009 with study visits taking place in 3 sites (The University of Chicago, Howard Brown Health Clinic, and the Respiratory Health Association). Follow-up interviews for the study concluded in April 2010.
Pre-assignment Details: * N=707 screened for participation (320 met exclusion criteria, 54/387 who passed chose not to participate)
  * 333 participants were randomized into the trial
Groups:
- Naltrexone - MALE: Males receiving naltrexone as part of the trial
- Placebo - MALE: Males receiving placebo as part of the trial
- Naltrexone - FEMALE: Females receiving naltrexone as part of the trial
- Placebo - FEMALE: Females receiving placebo as part of the trial
Period: Overall Study
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Started | 80 | 77 | 88 | 88
Received Study Treatment | 76 (n=4 did not start treatment (3 lost interest, 1 unknown)) | 71 (n=6 did not start treatment (1 diff treat. desired, 3 lost interest, 1 began psych meds, 1 unknown)) | 85 (n=3 did not start treatment (2 lost interest, 1 unknown)) | 83 (n=5 did not start treatment (2 health problems, 1 wanted diff. treatment method, 2 lost interest))
Completed | 58 (Discontinued: 1 smoking related, 1 reaction to tablet, 6 time commitment, 2 other, 8 unspecified) | 51 (Discontinued: 5 smoking related, 3 reaction to tablet, 2 time commitment, 1 other, 9 unspecified) | 65 (Discontinued: 5 smoking related, 4 reaction to tablet, 4 time commitment, 3 other, 4 unspecified) | 64 (Discontinued: 9 smoking related, 2 reaction to tablet, 4 time commitment, 1 other, 3 unspecified)
Not Completed | 22 | 26 | 23 | 24
Not completed — Lost Interest | 3 | 4 | 2 | 3
Not completed — Unknown/Unspecified | 11 | 11 | 8 | 4
Not completed — Protocol Violation | 1 | 6 | 5 | 11
Not completed — Unpleasant Reaction To Tablet | 1 | 3 | 4 | 2
Not completed — Time Commitment, Scheduling, or Travel | 6 | 2 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE | Total
Number analyzed (Participants) | 80 | 77 | 88 | 88 | 333
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 80 | 77 | 86 | 88 | 331
  >=65 years | 0 | 0 | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.45 (10.97) | 40.21 (10.98) | 44.34 (11.49) | 44.95 (10.45) | 42.13 (11.27)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 88 | 88 | 176
  Male | 80 | 77 | 0 | 0 | 157
Region of Enrollment [Number; unit: participants]
  United States | 80 | 77 | 88 | 88 | 333

OUTCOME MEASURES:

1. Primary Outcome: Prolonged Smoking Abstinence: 4 Weeks Post Quit-Date
Description: Prolonged Abstinence at 4 weeks post quit date (Study Week 7). Prolonged Abstinence defined as not smoking (even a puff of a cigarette) at any point during the previous time frame, allowing for a 1-week grace period.
Time Frame: 4 Weeks Following Smoking Quit Date (Study week 7)
Population: All participants who received study treatment by participating through smoking quit date (Study Week 3)were analyzed for this outcome.
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants | 43 | 29 | 40 | 39

2. Secondary Outcome: Weight Change at End of Treatment (Smoking Abstinent Only)
Description: Weight change in lbs at 12 weeks post smoking quit date (study week 15) for only those reporting continued smoking abstinence at the end of treatment. All data are Mean(SEM) and represent positive change, unless otherwise noted. Smoking abstinent for this measure defined as no smoking even 1 puff of a cigarette since the smoking quit date (study week 3), allowing for a 1-week grace period.
Time Frame: Weight change at 12 weeks post smoking quit date (study week 15)
Population: All participants completing through smoking quit date (study week 3) and who were smoking abstinent at end of treatment (study week 15)
Measure: Mean (Standard Error); unit: Pounds
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 23 | 12 | 17 | 23
Pounds | 4.79 (0.78) | 5.58 (0.78) | 2.26 (0.68) | 5.08 (0.69)

3. Primary Outcome: Prolonged Smoking Abstinence: 12 Weeks Post Quit-Date
Description: Prolonged Abstinence at 12 weeks post quit date (Study Week 15). Prolonged Abstinence defined as not smoking (even a puff of a cigarette) at any point during the previous time frame, allowing for a 1-week grace period.
Time Frame: 12 Weeks Following Smoking Quit Date (Study week 15)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants | 23 | 12 | 17 | 23

4. Primary Outcome: 7-Day Point Prevalence Smoking Abstinence: 4 Weeks Post Quit-Date
Description: 7-Day Point Prevalence smoking abstinence at 4 weeks post quit date (Study Week 7). 7-Day Point Prevalence abstinence defined as not smoking (even a puff) for seven days in a row or on one day in each of two consecutive weeks during the previous time frame.
Time Frame: 4 Weeks Following Smoking Quit Date (Study week 7)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants | 47 | 33 | 49 | 43

5. Secondary Outcome: Weight Change at End of Treatment (Regardless of Quit Status)
Description: Weight change at 12 weeks post quit date (study week 15) for the whole sample regardless of quit status. All data is Mean(SEM) and represents a positive change unless otherwise noted.
Time Frame: Weight change at 12 weeks post quit date (study week 15) from smoking quit date
Population: All participants who received study treatment by participating through smoking quit date (Study Week 3)were analyzed for this outcome, regardless of their abstinence status at 12 weeks post quit date (study week 15)
Measure: Mean (Standard Error); unit: Pounds
Groups:
- Placebo: Participants receiving Placebo as part of the trial
- Naltrexone: Participants receiving Naltrexone as part of the trial
Arm/Group | Placebo | Naltrexone
Number analyzed (Participants) | 154 | 161
Pounds | 5.29 (0.52) | 3.42 (0.53)

6. Primary Outcome: 7-Day Point Prevalence Smoking Abstinence: 12 Weeks Post Quit-Date
Description: 7-Day Point Prevalence smoking abstinence at 12 weeks post quit date (Study Week 15). 7-Day Point Prevalence abstinence defined as not smoking (even a puff) for seven days in a row or on one day in each of two consecutive weeks during the previous time frame.
Time Frame: 12 Weeks Following Smoking Quit Date (Study week 15)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants | 31 | 24 | 30 | 31

7. Primary Outcome: 7-Day Point Prevalence Smoking Abstinence: 26 Weeks Post Quit-Date
Description: 7-Day Point Prevalence smoking abstinence at 29 weeks post quit date (Study Week 29). 7-Day Point Prevalence abstinence defined as not smoking (even a puff) for seven days in a row or on one day in each of two consecutive weeks during the previous time frame.
Time Frame: 26 Weeks Following Smoking Quit Date (Study week 29)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants | 22 | 18 | 20 | 22

8. Primary Outcome: 7-Day Point Prevalence Smoking Abstinence: 52 Weeks Post Quit-Date
Description: 7-Day Point Prevalence smoking abstinence at 52 weeks post quit date (Study Week 55). 7-Day Point Prevalence abstinence defined as not smoking (even a puff) for seven days in a row or on one day in each of two consecutive weeks during the previous time frame.
Time Frame: 52 Weeks Following Smoking Quit Date (Study week 55)
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants | 14 | 15 | 14 | 20

9. Secondary Outcome: Opioid Antagonist Reported Side Effects: 1-Week Post Quit Date
Description: Participants reporting side effects during the previous week by pill type and sex, 1-week following quit date (Study week 4). Participants rated side effects experienced by None, Mild, or Severe.
Time Frame: 1-Week Post Quit Date (Study Week 4)
Population: All participants who received study treatment by participating through smoking quit date (Study Week 3) were analyzed for this outcome.
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants
  Nausea - "Mild" | 16 | 5 | 24 | 13
  Nausea - "Severe" | 4 | 3 | 4 | 2
  Vomiting - "Mild" | 3 | 0 | 3 | 5
  Vomiting - "Severe" | 1 | 0 | 2 | 0
  Headache- "Mild" | 28 | 17 | 31 | 33
  Headache - "Severe" | 4 | 2 | 0 | 2
  Light Headed/Dizzy - "Mild" | 22 | 16 | 25 | 17
  Light Headed/Dizzy - "Severe" | 5 | 1 | 1 | 0
  Flushed/Warm - "Mild" | 12 | 9 | 24 | 15
  Flushed/Warm - "Severe" | 1 | 1 | 6 | 6
  Tiredness - "Mild" | 42 | 34 | 38 | 33
  Tiredness - "Severe" | 5 | 7 | 10 | 9
  Anxiety/Agitation - "Mild" | 33 | 35 | 31 | 32
  Anxiety/Agitation - "Severe" | 3 | 3 | 3 | 6
  Increased Sexual Desire - "Mild" | 10 | 22 | 9 | 6
  Increased Sexual Desire - "Severe" | 2 | 6 | 1 | 0
  Insomnia - "Mild" | 13 | 16 | 19 | 12
  Insomnia - "Severe" | 2 | 3 | 5 | 3
  Constipation - "Mild" | 18 | 20 | 24 | 14
  Constipation - "Severe" | 1 | 1 | 1 | 3
  Diarrhea - "Mild" | 6 | 6 | 5 | 7
  Diarrhea - "Severe" | 2 | 0 | 0 | 1
  Joint or Muscle Pain - "Mild" | 21 | 21 | 14 | 13
  Joint or Muscle Pain - "Severe" | 0 | 2 | 2 | 5

10. Secondary Outcome: Opioid Antagonist Reported Side Effects: 4-Weeks Post Quit Date
Description: Participants reporting side effects during the previous week by pill type and sex, 4-weeks following quit date (Study week 7). Participants rated side effects experienced by None, Mild, or Severe.
Time Frame: 4-Weeks Post Quit Date (Study Week 7)
Population: as for outcome 9
Measure: Number; unit: Participants
Arm/Group | Naltrexone - MALE | Placebo - MALE | Naltrexone - FEMALE | Placebo - FEMALE
Number analyzed (Participants) | 76 | 71 | 85 | 83
Participants
  Nausea - "Mild" | 3 | 3 | 12 | 7
  Nausea - "Severe" | 3 | 1 | 0 | 0
  Vomiting - "Mild" | 1 | 0 | 1 | 0
  Vomiting - "Severe" | 0 | 0 | 0 | 0
  Headache- "Mild" | 18 | 23 | 19 | 19
  Headache - "Severe" | 3 | 1 | 2 | 1
  Light Headed/Dizzy - "Mild" | 11 | 7 | 17 | 14
  Light Headed/Dizzy - "Severe" | 2 | 0 | 1 | 0
  Flushed/Warm - "Mild" | 6 | 5 | 22 | 14
  Flushed/Warm - "Severe" | 0 | 2 | 3 | 1
  Tiredness - "Mild" | 27 | 27 | 32 | 24
  Tiredness - "Severe" | 2 | 2 | 7 | 7
  Anxiety/Agitation - "Mild" | 18 | 19 | 27 | 23
  Anxiety/Agitation - "Severe" | 2 | 3 | 4 | 3
  Increased Sexual Desire - "Mild" | 25 | 17 | 11 | 7
  Increased Sexual Desire - "Severe" | 2 | 4 | 1 | 2
  Insomnia - "Mild" | 10 | 13 | 17 | 10
  Insomnia - "Severe" | 1 | 1 | 1 | 2
  Constipation - "Mild" | 13 | 8 | 18 | 10
  Constipation - "Severe" | 2 | 2 | 2 | 1
  Diarrhea - "Mild" | 7 | 11 | 6 | 4
  Diarrhea - "Severe" | 2 | 0 | 0 | 1
  Joint or Muscle Pain - "Mild" | 17 | 15 | 15 | 16
  Joint or Muscle Pain - "Severe" | 2 | 2 | 1 | 1

ADVERSE EVENTS:
Description: Number of participant at risk represent those assigned to either Naltrexone or Placebo condition (i.e. receiving treatment) - Placebo: n=154, Naltrexone: n=161
Arm/Group | Placebo | Naltrexone
Serious Adverse Events (participants affected / at risk) | 2/154 | 2/161
Other Adverse Events (participants affected / at risk) | 92/154 | 101/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=154) | Naltrexone (N=161)
Benign Brain Mass (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) — Participant reported this during time of study; however, diagnosed as having developed prior to study participation
Suicidal Ideation Remitting in 2 Days with Recurrence (Psychiatric disorders) | 0 (0) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Motor Vehicle Collision (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=154) | Naltrexone (N=161)
Nausea (General disorders) | 26 | 52
Vomiting (General disorders) | 5 | 10
Headache (General disorders) | 57 | 67
Lightheaded or dizzy (General disorders) | 37 | 57
Flushed or warm (General disorders) | 36 | 46
Tiredness (General disorders) | 91 | 98
Agitation or anxiety (General disorders) | 82 | 76
Increased Sexual Desire (General disorders) | 37 | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No